CLINICAL TRIAL: NCT02628860
Title: Efficacy of Ferric Carboxymaltose (Ferinject®) in Anemic Patients Anticipating Pancreatoduodenectomy
Acronym: FCM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: JW Pharmaceutical (Industry)
Responsible Party: Principal Investigator, Sang-Jae Park, Head of Center for Liver Cancer, Chief of the Liver and Pancreatobiliary Cancer Branch, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-13-709
Record Dates: First submitted 2015-02-05; First posted 2015-12-11 (Estimated); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Pancreatic Cancer; Anemia
Keywords: ferric carboxymaltose; Ferinject®; pancreatoduodenectomy
MeSH Terms: conditions — Pancreatic Neoplasms; Anemia | interventions — ferric carboxymaltose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ferinject (Experimental): Ferinject to be administered as IV drip infusion or undiluted bolus injection with a minimum administration time of 15minutes (for 1000mg single administration) for body weight ≥50 Kg or 6 minutes (for 500mg single administration) for body weight <50 Kg .
  Dosage form: 5% w/v iron containing 50 mg iron per mL, as sterile solution of FERINJECT® in water for injection. In case of drip infusion FERINJECT® must be diluted only in sterile 0.9% sodium chloride.
  Strength/Packaging: 10 mL vials containing 500 mg iron as iron per vial.
  Interventions: Drug: Ferinject (Ferric Carboxymaltose)

INTERVENTIONS:
Drug: Ferinject (Ferric Carboxymaltose) — Ferinject® to be administered as IV drip infusion or undiluted bolus injection with a minimum administration time of 15minutes (for 1000mg single administration) for body weight ≥50 Kg or 6 minutes (for 500mg single administration) for body weight <50 Kg .
  Study drug may be administered as IV drip infusion or IV undiluted bolus injection.
  Other Names: Ferinject

SUMMARY:
This phase II study is to evaluate the safety and efficacy of Ferinject® in reducing perioperative transfusion in iron deficiency anemia patients anticipating pancreatoduodenectomy.

DETAILED DESCRIPTION:
Primary objectives : Perioperative transfusion rate (including preop, intraop, postop≦7 days).

Secondary objectives : Postoperative complication, hospital stay, change of hematological parameters (Hb, ferritin, transferrin saturation (TSAT) change after Ferinject® injection), adverse effect with Ferinject® injection.

ELIGIBILITY:
Inclusion Criteria:

* ≥19 years old
* anticipating PD
* preoperative Hb of Female 7.0-11.9g/dl and Male 7.0-12.9g/dl
* signed written informed consent

Exclusion Criteria:

* a concurrent medical condition(s) that would prevent compliance or participation or jeopardize the health of the patient
* hypersensitivity to any component of the formulation
* active severe infection/inflammation
* history of transfusion, erythropoietin, >500 mg intravenous iron administration within 4 weeks prior to screening.
* history of acquired iron overload.
* MCV > 95µm3 or TSAT > 35%
* patients with preoperative Hb<7 g/dl
* pregnancy or lactation
* decreased renal function (defined as creatinine clearance <50 L/min/1.73m2calculated by eGFR(MDRD))
* chronic liver disease or increase of liver enzymes (ALT, AST) >5 times the upper limit of normal range

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-01; Primary Completion 2020-04-27 (Actual); Study Completion 2020-04-27 (Actual)

PRIMARY OUTCOMES:
Perioperative transfusion rate | from preoperative baseline within the first 7 days after surgery
  To evaluate reducing transfusion rate during perioperative period

SECONDARY OUTCOMES:
Assessment of complications after surgery as assessed by Clavien-Dindo classification of surgical complications | up to 4-6 weeks after surgery
  To investigate the association between the number of participants with complications and hospital length of stay(days)
Change of hematology parameters | up to 4-6 weeks after surgery
  change of hematology parameters value of Hb in g/dL,
  * ferritin in ng/ml
  * transferrin saturation in % (TSAT) after Ferinject® administration)
Adverse event | up to 4-6 weeks after surgery
  assessment of adverse effect with Ferinject® administration

CONTACTS AND LOCATIONS:
Overall Officials: Sang Jae Park, M.D, Principal Investigator — Study Principal Investigator
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Park SJ, Kim SW, Jang JY, Lee KU, Park YH. Intraoperative transfusion: is it a real prognostic factor of periampullary cancer following pancreatoduodenectomy? World J Surg. 2002 Apr;26(4):487-92. doi: 10.1007/s00268-001-0254-6. Epub 2002 Feb 4. PMID 11910485
- [Result] Yeh JJ, Gonen M, Tomlinson JS, Idrees K, Brennan MF, Fong Y. Effect of blood transfusion on outcome after pancreaticoduodenectomy for exocrine tumour of the pancreas. Br J Surg. 2007 Apr;94(4):466-72. doi: 10.1002/bjs.5488. PMID 17330243
- [Result] Peters JH, Carey LC. Historical review of pancreaticoduodenectomy. Am J Surg. 1991 Feb;161(2):219-25. doi: 10.1016/0002-9610(91)91134-5. PMID 1990875
- [Result] Kaplan J, Sarnaik S, Gitlin J, Lusher J. Diminished helper/suppressor lymphocyte ratios and natural killer activity in recipients of repeated blood transfusions. Blood. 1984 Jul;64(1):308-10. PMID 6234037
- [Result] Waymack JP, Gallon L, Barcelli U, Trocki O, Alexander JW. Effect of blood transfusions on immune function. III. Alterations in macrophage arachidonic acid metabolism. Arch Surg. 1987 Jan;122(1):56-60. doi: 10.1001/archsurg.1987.01400130062009. PMID 3492188
- [Result] Innerhofer P, Tilz G, Fuchs D, Luz G, Hobisch-Hagen P, Schobersberger W, Nussbaumer W, Lochs A, Irschick E. Immunologic changes after transfusion of autologous or allogeneic buffy coat-poor versus WBC-reduced blood transfusions in patients undergoing arthroplasty. II. Activation of T cells, macrophages, and cell-mediated lympholysis. Transfusion. 2000 Jul;40(7):821-7. doi: 10.1046/j.1537-2995.2000.40070821.x. PMID 10924610
- [Result] Ghio M, Contini P, Mazzei C, Brenci S, Barberis G, Filaci G, Indiveri F, Puppo F. Soluble HLA class I, HLA class II, and Fas ligand in blood components: a possible key to explain the immunomodulatory effects of allogeneic blood transfusions. Blood. 1999 Mar 1;93(5):1770-7. PMID 10029607
- [Result] Burrows L, Tartter P. Effect of blood transfusions on colonic malignancy recurrent rate. Lancet. 1982 Sep 18;2(8299):662. doi: 10.1016/s0140-6736(82)92764-7. No abstract available. PMID 6125797
- [Result] Griffin JF, Smalley SR, Jewell W, Paradelo JC, Reymond RD, Hassanein RE, Evans RG. Patterns of failure after curative resection of pancreatic carcinoma. Cancer. 1990 Jul 1;66(1):56-61. doi: 10.1002/1097-0142(19900701)66:13.0.co;2-6. PMID 2354408